CLINICAL TRIAL: NCT01017380
Title: Comparing Etoricoxib and Celecoxib for Preemptive Analgesia for Acute Postoperative Pain in Patients Undergoing Arthroscopic Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial
Brief Title: Preemptive Analgesia in Cruciate Reconstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Secretariate,Department of Orthopaedic Surgery, Facuty of Medicine, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC50/369-007
Record Dates: First submitted 2009-11-17; First posted 2009-11-20 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: preemptive analgesia; cruciate ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Celecoxib; Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- placebo (Experimental): identical placebo
  Interventions: Drug: Celecoxib; Drug: etoricoxib

INTERVENTIONS:
Drug: Celecoxib — celecoxib 400 mg 1 cap before surgery
Drug: etoricoxib — 120 mg 1 tab before surgery

SUMMARY:
The aims of this study was to compare analgesic efficacy of preoperative administration of etoricoxib versus celecoxib for post-operative pain relief after arthroscopic anterior cruciate ligament reconstruction. One hundred and two patients diagnosed as anterior cruciate ligament injury will randomized into 3 groups using opaque envelope. Both patients and surgeon were blinded to the allocation. All of the patients will be operated by one orthopaedic surgeon under regional anesthesia. Each group will be given either etoricoxib 120 mg., celecoxib 400 mg., or placebo 1 hour prior to operative incision. Post-operative pain intensity, time to first dose of analgesic requirement and numbers of analgesic used for rescue pain control and adverse events will be recorded periodically to 48 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients with anterior cruciate ligament injury age 15-50 yr

Exclusion Criteria:

* previous knee surgery

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
VAS score | 6,12,24,48 hour postoperative

SECONDARY OUTCOMES:
number of analgesic used | 48 hour postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Boonsin Tangtrakulwanich, MD.,Ph.D, Study Director — Faculty of Medicine, Prince of Songkla University
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

REFERENCES:
- [Derived] Boonriong T, Tangtrakulwanich B, Glabglay P, Nimmaanrat S. Comparing etoricoxib and celecoxib for preemptive analgesia for acute postoperative pain in patients undergoing arthroscopic anterior cruciate ligament reconstruction: a randomized controlled trial. BMC Musculoskelet Disord. 2010 Oct 25;11:246. doi: 10.1186/1471-2474-11-246. PMID 20973952